CLINICAL TRIAL: NCT04470557
Title: The Relationship Between Lab Finding and COVID-19 Severity: Multicenter Study
Brief Title: Relation Between Lab Finding and COVID-19 Severity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Anwar Mohamed Ali, principal investigator, Assiut University
Other Study IDs: RLCS
Record Dates: First submitted 2020-07-11; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: Laboratory; Severity; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COVID-19: The patients will be subjected to to laboratory analyses, a number of hematological, immunological and biochemical parameters like total leucocytic count and differential count of CBC, ESR, D- dimer levels in plasma, CRP, serum urea and creatinine levels, serum levels of AST, ALT liver enzymes, serum ferritin levels Also, CT scan of chest, clinical assessment and the severity and course of the disease.
  Interventions: Diagnostic Test: D-dimer,CBC.ESR,CRP,; Diagnostic Test: Liver function tests ,serum ferritin and PCR for COVID-19 .

INTERVENTIONS:
Diagnostic Test: D-dimer,CBC.ESR,CRP, — Complete blood count (for patients and control subjects): was done on CELL-DYN 3700 (Abbott-Germany) and blood film was stained by leishman staining, the morphology of red blood cells. CRP titre estimation by latix method .ESR erythrocyte sedimentation rate estimation (1:5) by Westerngreen tube method.
Diagnostic Test: Liver function tests ,serum ferritin and PCR for COVID-19 . — Serum ferritin was performed for all subjects on Modular P auto analyzer (Roche Diagnostics, Mannheim, Germany),
  • Liver function tests ( aspartate aminotransferase, alanine aminotransferase and alkaline phosphatase) and kidney funcrion were performed for all subjects on Modular P auto analyzer (Roche Diagnostics, Mannheim, G ermany),

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (COVID-19) poses substantial challenges for health care systems. With a vastly expanding amount of publications on COVID-19, clinicians need evidence synthesis to produce guidance for handling patients with COVID-19.

DETAILED DESCRIPTION:
. Conavirus belongs to the subfamily of Ortho-coronavirinae in the family of Coronaviridae and the Order Nidovirales. In 2003, a SARS-CoV had caused the out- break of severe acute respiratory syndrome. In December 2019, an "unknown viral pneumonia" out- break has been reported. Finally, a novel coronavirus was detected, isolated virus was termed as SARS-CoV2, characterized as highly contagious and deadly. By the end of February 2020, more than 78,631 cases infected with SARS-CoV-2, and more than 2747 deaths were confrmed in China, and the COVID-19 has been declared a pan- demic by World Health Organization. For those infected by SARS-CoV-2, some of the patients didnot show hypoxemia or respiratory stress during the course of COVID-19, indicating a multifaceted disease of SARS-CoV-2 infection. Therefore, one reliable and convenient biomarker is needed to predict the severity of COVID-19 pneumonia. Recently, several studies have reported that C-reactive protein (CRP) is positively asso-ciated with severe dengue infection, and patients with higher plasma CRP in the initial period of dengue, are at higher risk to develop plasma leakage. We examined which routine laboratory tests are associated with severe COVID-19 disease, and the relation between the laboratory results and the security of COVID19 diasease, in two of large Upper Egypt medical centers, which are Aswan University and assiut university hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Age: all ages.
* Sex: Males and females.
* COVID-19 patients approved by positive PCR.

Exclusion Criteria:

* Patients with known chronic chest disease preceding the infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted on 100 patients with COVID-19 patients of all age groups and both sexes.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of severity of patients with COVID-19 in relation to Laboratory findings. | up to 1 month
  with successful completion of the aim, the investigators will establish the correlation between laboratory findings and severity of COVID-19 patients according to WHO classification.

CONTACTS AND LOCATIONS:
Overall Officials: Esam_eldeen M. Abdalla, Doctorate, Study Chair — Assiut University; Heba Abdellatif, Doctorate, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Du RH, Li B, Zheng XS, Yang XL, Hu B, Wang YY, Xiao GF, Yan B, Shi ZL, Zhou P. Molecular and serological investigation of 2019-nCoV infected patients: implication of multiple shedding routes. Emerg Microbes Infect. 2020 Feb 17;9(1):386-389. doi: 10.1080/22221751.2020.1729071. eCollection 2020. PMID 32065057
- [Background] Chen CC, Lee IK, Liu JW, Huang SY, Wang L. Utility of C-Reactive Protein Levels for Early Prediction of Dengue Severity in Adults. Biomed Res Int. 2015;2015:936062. doi: 10.1155/2015/936062. Epub 2015 Jul 12. PMID 26247033
- [Result] Alnor A, Sandberg MB, Gils C, Vinholt PJ. Laboratory Tests and Outcome for Patients with Coronavirus Disease 2019: A Systematic Review and Meta-Analysis. J Appl Lab Med. 2020 Sep 1;5(5):1038-1049. doi: 10.1093/jalm/jfaa098. PMID 32573713